CLINICAL TRIAL: NCT03376646
Title: A Multicenter, Randomized, Controlled Clinical Study to Evaluate the Efficacy and Safety of Dissolve™ Compared to Resolute™ Integrity in Treatment of Coronary Small Vessel Disease in Chinese Population
Brief Title: A Safety and Efficacy Study of Dissolve™ in Treatment of Coronary Small Vessel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DK Medical Technology (Suzhou) Co., Ltd. (Industry)
Collaborators: Core Medical (Beijing) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-VP-02
Record Dates: First submitted 2017-12-08; First posted 2017-12-18 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Coronary Small Vessel Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A: Dissolve™ (Experimental)
  Interventions: Device: Cohort A: Dissolve™
- Cohort A: Resolute™ Integrity (Active Comparator)
  Interventions: Device: Cohort A: Resolute™ Integrity
- Cohort B: Dissolve™-2.00mm (Experimental): Cohort B is single arm.
  Interventions: Device: Cohort B: Dissolve™-2.00mm

INTERVENTIONS:
Device: Cohort A: Dissolve™ — Dissolve™ are to be used in the trial
  Other Names: Paclitaxel coated balloon
  Arms: Cohort A: Dissolve™
Device: Cohort A: Resolute™ Integrity — Resolute™ Integrity are to be used in the trial
  Other Names: Zotarolimus eluting stent
  Arms: Cohort A: Resolute™ Integrity
Device: Cohort B: Dissolve™-2.00mm — Dissolve™ are to be used in the trial
  Arms: Cohort B: Dissolve™-2.00mm

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety in the treatment of Coronary Small Vessel Disease by drug coated balloon (DCB) Dissolve™ versus drug eluting stent (DES) Resolute™ Integrity.

ELIGIBILITY:
Inclusion Criteria:

Related to the patients:

Cohort A:

1. Patients who agree to accept the angiography follow-up visit at 9-month and follow up visits at 1-month, 6-month, 9-month, 1-year, 2-year, 3-year, 4-year and 5-year
2. Patients with stable angina, unstable angina, old myocardial infarction (including ST elevation MI or Non-ST elevation MI) or proven asymptomatic ischemia
3. Patients who can receive any kind of coronary revascularization (including balloon angioplasty, stent implantation or coronary artery bypass grafting)

   Cohort B: All candidates for Cohort B of this study must meet number 1, 2 of the above criteria and
4. Patients who can receive balloon angioplasty

   Related to lesion:

   Cohort A
5. The reference blood vessel diameter is 2.25 mm-2.75 mm, length ≤ 26mm
6. Before surgery, stenosis diameter must be ≥ 70% or ≥ 50% and accompanied by ischemia
7. One subject is allowed to have 1 target lesion at most (Two lesions can be treat as one target lesion, if they are in the same vessel, with the distance less than 10mm, with total length ≤ 26mm, and can be intervened by one DCB or DES)

   Cohort B: All candidates for Cohort B of this study must meet number 6,7 of the above criteria and
8. The reference blood vessel diameter is 2.00mm-2.25mm

Exclusion Criteria:

Related to patients

1. Patients who had Myocardial Infarction within 1 week before being included
2. Patients with severe congestive heart failure or NYHA grade IV heart failure
3. Left ventricular ejection fraction (LVEF) < 35%
4. Patients who had heart transplantation
5. Patients with severe valvular heart disease
6. The patients had cerebral stroke within 6 months before being included, or have a history of peptic ulcer or gastrointestinal bleeding, or the patients have a bleeding tendency according to the investigator
7. Patients with leukopenia (white blood cell count < 3×10^9/L) for more than three days; Patients with low neutrophil counts (ANC < 1000/mm^3) for more than three days; Patients with thrombocytopenia (platelet count < 100,000/mm^3)
8. Patients with renal insufficiency (eGFR < 30mL/min)
9. Patients who are forbidden to use anticoagulation agents or anti-platelet drugs, and unable to tolerate Aspirin or Clopidogrel
10. Patients who are allergic to Paclitaxel or Zotarolimus
11. The patients have a life expectancy of less than 12 months, or it would be difficult to finish follow-ups within 12 months
12. Pregnant or lactating women, or women who plan to get pregnant within 12 months or refuse to take effective contraceptives
13. The patients are participating in any other clinical trials before reaching the primary endpoints
14. Patients who are unsuitable for the study according to the investigator due to other reasons

    Related to the Lesion:
15. Patients with total occlusion at the target lesion
16. Patients who have severe calcification of the target lesion, and balloon pre-dilatation could not be performed successfully
17. The target lesions are bifurcation lesion with the diameter of the branch vessel > 2.00mm
18. The target lesions are in-stent restenosis
19. Angiography indicates thrombosis in the target vessel
20. Complicated with lesions in left main (LM) coronary requiring intervention treatment
21. More than 2 non-target lesions need treatment, or the non-target lesion could not be intervened successfully before the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
In-segment percent diameter stenosis of the target lesion at 9 months after procedure | 9 months after the procedure

SECONDARY OUTCOMES:
Device success rate of the interventional therapy | From the start of index procedure to the end of index procedure, Day 0
  Successful delivery and use of the assigned balloon/stent at the intended target lesion and successful withdrawal of the delivery system with attainment of final residual stenosis of less than 50% and TIMI 3 blood flow (DCB arm) or less than 30% and TIMI 3 blood flow (DES arm) by visual estimation
Lesion success rate of the interventional therapy | From the start of index procedure to the end of index procedure, Day 0
  Attainment of final residual stenosis of less than 50% and TIMI 3 blood flow (DCB arm) or less than 30% and TIMI 3 blood flow (DES arm) by visual estimation.
Clinical success rate of the interventional therapy | 7 days after the procedure
  Without the occurrence of cardiac death, target vessel Myocardial Infarction (MI) or repeat target lesion revascularization (TLR).
In-device percent diameter stenosis of the target lesion | 9 months after the procedure
  Restenosis is defined as stenosis > 50% by angiography
In-device minimal lumen diameter (MLD) | 9 months after the procedure
In-segment MLD | 9 months after the procedure
In-device late lumen loss (LLL) | 9 months after the procedure
In-segment LLL | 9 months after the procedure
Binary restenosis rate in lesion section | 9 months after the procedure
Target vessel revascularization (TVR) rate | 1 month, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years after the procedure
Target lesion failure (TLF) rate | 1 month, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years after the procedure
Target lesion revascularization (TLR) rate | 1 month, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years after the procedure
Rate of all adverse events and severe adverse events | 1 month, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years after the procedure
Rate of major adverse cardiovascular events | 1 month, 6 months, 9 months, 1 year, 2 years, 3 years, 4 years and 5 years after the procedure
  Including death, myocardial infarction (MI), stroke and renal failure

CONTACTS AND LOCATIONS:
Overall Officials: Shubin Qiao, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (15):
- China (15):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Hospital, Beijing
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University People's Hospital, Capital Medical University, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital of Dalian Medical University, Dalian
  - The Second Affiliated Hospital of Dalian Medical University, Dalian
  - General Hospital of Daqing Oil Field, Daqing
  - Sir Run Run Shaw Hospital, Zhejiang University School of medicine, Hangzhou
  - Union Hospital, Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - General Hospital of Ningxia Medical University, Yinchuan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu S, Zhou Y, Shen Z, Chen H, Qiu C, Fu G, Li H, Yu Z, Zeng Q, Li Z, Li W, Qiao S; Dissolve SVD investigators. Comparison of Drug-Coated Balloon and Drug-Eluting Stent for the Treatment of Small Vessel Disease (from the Dissolve SVD Randomized Trial). Am J Cardiol. 2024 Jan 15;211:29-39. doi: 10.1016/j.amjcard.2023.05.057. Epub 2023 Nov 22. PMID 37995506